CLINICAL TRIAL: NCT00871624
Title: Efficacy and Safety of Dexmedetomidine During Non-Invasive Positive Pressure Ventilation for Patients With Acute Respiratory Failure: A Randomized, Double-blind, Placebo-controlled Pilot Study
Brief Title: Efficacy and Safety of Dexmedetomidine During Non-Invasive Positive Pressure Ventilation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TuftsMedicalCenter 8533
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Subjects received active dexmedetomidine 0.2 -0.7 mcg/kg/hr
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Subjects received placebo saline solution 0.2-0.7 mcg/kg/hr
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be started at a rate of 0.2mcg/kg/hr and titrated by 0.1 mcg/kg/hr every 30 minutes to a maximum of 0.7 mcg/kg/hr to maintain a Riker-SAS 3-4.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Placebo — Placebo infusion will be started at a rate of 0.2mcg/kg/hr and titrated by 0.1 mcg/kg/hr every 30 minutes to a maximum of 0.7 mcg/kg/hr to maintain a Riker-SAS 3-4.
  Other Names: Precedex
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the efficacy and safety of dexmedetomidine during Non-invasive positive pressure ventilation (NPPV) for patients with acute respiratory failure compared to standard analgesic/sedation practices

DETAILED DESCRIPTION:
Non-invasive positive-pressure ventilation (NPPV) is increasingly being used to manage patients with acute respiratory failure (ARF) in an effort to avoid the numerous negative sequelae associated with intubation and mechanical ventilation. In the USA, it is estimated that 20-30% of all patients placed on mechanical ventilation are treated with NPPV. Indications for NPPV include but are not limited to acute or acute-on-chronic hypercapnic respiratory failure, pulmonary edema, respiratory failure in immunocompromised patients or that due to chest wall deformity or neuromuscular disease. For NPPV to be successful, it is critical that the patient be cooperative and comfortable (i.e. no pain) as agitation and discomfort interfere with the success of NPPV.

Despite the importance of patient comfort during NPPV, physicians infrequently use sedation or analgesic therapy during NPPV, primarily due to concerns about the respiratory depressant effects of most of the sedatives (e.g., benzodiazepines) and analgesics (e.g., opioids) that are currently available. In addition, neither the benzodiazepines nor opioids are easily titratable, can easily accumulate and can be associated with both the development of delirium and a withdrawal effect.

Dexmedetomidine is an intravenous rapid-onset, short acting ά 2-receptor agonist that is approved for short-term sedation in post-operative and critically ill patients. It has been stated that this drug produces a state of "cooperative sedation" allowing the patient to interact with health care providers. Dexmedetomidine has been used for its ability to cause sympatholysis and, because of analgesic properties, to decrease the need for opioids. Potential advantages include its short half life and intravenous route of administration, permitting rapid titration to achieve sedation targets and, in patients with respiratory failure; it can provide both sedation and analgesia without inducing respiratory depression. Despite these advantages, it is currently used by less than 5% of pulmonologists/ intensivists as the primary sedative option during NPPV and has not been studied in a controlled fashion in this population. Therefore, dexmedetomidine may prove to be more efficacious and safe compared to standard sedation/analgesic therapy during NPPV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute respiratory failure requiring the initiation of NPPV
* Admission to the medical ICU service at Tufts Medical Center or Winchester Hospital

Exclusion Criteria:

* Patients with delirium (intensive care delirium screening checklist score ≥ 4) or disorientation (not oriented to person or place)
* Receiving NPPV for ≥ 8 hours (includes treatment with NPPV at an outside hospital)
* Intubation and mechanical ventilation in the past month based on hospital admission note
* Age ≥ 85 years
* Inability of the potential subject to give informed consent
* Current treatment with antipsychotic agent based on hospital admission note
* Heart rate ≤ 50 bpm
* Systolic blood pressure ≤ 90 mmHg
* History of heart block without pacemaker use or severe ventricular dysfunction (EF ≤25%) based on hospital admission note
* Acute alcohol withdrawal based on hospital admission note
* History of end stage liver failure (based on presence of ≥ 1 or more of the following: AST/ALT ≥ 2 times ULN, INR ≥ 2, total bilirubin ≥ 1.5
* Irreversible brain disease consistent with severe dementia based on hospital admission note
* Pregnancy (all women of child-bearing age will undergo a pregnancy test prior to study enrollment)
* Treatment with clonidine or dexmedetomidine in the past 30 days based on hospital admission note
* Known allergy or sensitivity to clonidine or dexmedetomidine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Principal Investigator — Tufts Medical Center / Winchester Hospital
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 18 | 18
Completed | 16 | 17
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6) | 62 (17) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of NIV as Assessed by an NIV Tolerance Score
Description: NIV tolerance (NIV intolerance score =1 out of 4) A score of 1 for a comfortable and relaxed patient tolerating NIV; a score of 2 for mild intolerance with some discomfort and occasionally grabbing at the NIV mask; a score of 3 for moderate intolerance and discomfort with the NIV mask most of the time but more frequent grabbing at the mask, sometimes pulling it off; and a score of 4 for severe NIV intolerance with agitation and the inability to leave the NIV mask in place. The outcome measure description of the time frame is reported as the average of the NIV tolerance scores reported at the various time frames (0min, 30min, 60 min, 3hr, 6hr, 12hr, and then every 12hr after the start of NIV therapy up to 72 hours)
Time Frame: Completed at time 0min, 30min, 60min, 3hr, 6hr, 12hr, and then every 12 hours after the start of NPPV therapy up to 72 hours
Measure: Median (Inter-Quartile Range); unit: percentage of time spent tolerant to NIV
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 16 | 17
percentage of time spent tolerant to NIV | 99 [61 to 100] | 67 [40 to 100]
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Test type: Non-Inferiority or Equivalence — A difference in the mean four-point NIV intolerance score of 1 over the course of the study or between groups was considered through investigator consensus to be clinically meaningful. Assuming that the SD of NIV intolerance scores was 1 and that an alpha of 0.05 would be used for testing, it was determined that 18 subjects were needed in each group to achieve an 80% power; p = 0.54, Chi-squared; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.44 to 4.7]

2. Secondary Outcome: Percent of Study Time Spent With a Riker-SAS Score Between 3 and 4 Inclusive
Description: Percentage of time spent at desired sedation goal
Time Frame: Completed at baseline and every 4 hours after the start of NPPV therapy for the duration of the study
Measure: Median (95% Confidence Interval); unit: percentage of time
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 16 | 17
percentage of time | 100 [86 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Dexmedetomidine vs Placebo; Test type: Other; p = 0.3, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected hourly/daily throughout the study period
Arm/Group | Dexmedetomidine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No